CLINICAL TRIAL: NCT06881368
Title: Phenotypic and Etiological Characterization of Susac Syndrome
Acronym: CARESS Cohorte
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241173; 2025-A00214-45 (Other: ANSM ID-RCB)
Record Dates: First submitted 2025-01-29; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Susac Syndrome
MeSH Terms: conditions — Susac Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
SUSAC's Syndrome (SS) is characterized by the clinical triad of encephalopathy, hearing loss, and retinal artery branch occlusions. Since the first description of SS in 1979, hundreds of patients with SS, mostly young women, have been reported. However, comprehensive epidemiological, clinical and etiological features of SS have never been specifically addressed so far.

DETAILED DESCRIPTION:
Susac's Syndrome (SS) is characterized by the clinical triad of encephalopathy, hearing loss, and retinal artery branch occlusions. Since the first description of SS in 1979, hundreds of patients with SS, mostly young women, have been reported. However, comprehensive epidemiological, clinical and etiological features of SS have never been specifically addressed so far.

The diagnosis of SS is difficult because its characteristic signs often do not occur simultaneously or may be too subtle for the patient to notice. Neurological features of SS may occur several months prior to other symptoms. The retinal artery branch occlusion, by occurring in the peripheral portion of the retina, may remain asymptomatic. Sensorineural hearing loss may also be asymptomatic and disclosed only by audiogram. Besides mild pleocytosis in cerebro-spinal fluid, all performed biological tests are virtually negative. No infectious agent, consistent autoimmune marker, or coagulopathy has been disclosed. Changes seen on brain MRI are well characterized although not specific. The only site from which biopsy material is available for pathological analysis is the brain. The most common finding in brain biopsies is the presence of microinfarcts but brain biopsy is not currently performed.

Although the treatment of SS has not been studied in controlled trials, most patients have a good response to treatment with glucocorticoids, with the addition of antithrobomtic therapy and, for cases in which the disease is refractory to steroids, intravenous immune globulin or cyclophosphamide. The clinical course is characterized by recurrent attacks involving 1 or more components of the triad that characterize the active phase of the disease. Remission usually occurs after the active phase but some patients show residual mild to moderate dementia or gait disturbance, and impaired hearing and vision.

Susac's Syndrome is a vasculopathy causing small infarcts in the cochlea, retina and brain. Proposed explanations include a hypercoagulable state, vasospasm, and vasculitis, none of which are supported by laboratory results or findings on brain biopsies. The unique distribution of arteriolar disease affecting the brain, the retina, and the cochlea suggests selective vulnerability of these three structures. The brain, retina, and cochlea all have a blood-tissue barrier, and the endothelium in these sites shares a common embryologic origin and unique structural and antigenic characteristics. It has therefore been proposed that SS is an autoimmune disease in which the endothelium is the primary target, and damage to the endothelium triggers arteriolar occlusion and microinfarcts. However, the pathogenesis remains unknown.

The objective of this study is to characterize the epidemiological, clinical, and etiological features of Susac's Syndrome. In this aim, we will constitute a national clinical-based cohort including all SS new cases prospectively observed. French Society of Neurology, Ophtalmology and Internal Medicine will be asked to collaborate.The exhaustive and systematic analysis of each case will help to better define different aspects of the disease such as the incidence and prevalence, the clinical presentation, the diagnostic modalities and the impact of treatments.

Because Susac's syndrome is a rare disease, we expect to include 180 patients in this cohort. The constitution of the cohort will last for 9 years.

The conclusion of the study, based on statistical analysis done once all patients will be included in the cohort, should allow new recommendations in the diagnosis strategy and give new understandings of the therapeutic management of the disease. The result of this study may also give rise to hypothesis for an interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient presenting with at least two of the signs of the clinical triad: encephalopathy, cochlear damage authenticated by an audiogram (uni- or bilateral, predominantly in the middle or low frequencies), retinal artery occlusion assessed by fundoscopy or fluorescein retinal angiography.

Exclusion Criteria:

* Patient having been individually informed and objecting to the use of his/her data
* Patient under legal protection (guardianship or curatorship)
* Differential diagnosis established: multiple sclerosis, mitochondriopathy, CADASIL, primary tumour of the central nervous system, Lyme disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be studied will be patients with defined Susac syndrome, presenting with at least two of the signs of the clinical triad, having compatible complementary examinations and after elimination of differential diagnoses (see inclusion and non-inclusion criteria below). Patients will be included prospectively.
  The existence of an associated pathology (autoimmune, tumour, metabolic, etc.) is not a criterion for exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2037-03-30 (Estimated); Study Completion 2038-03-30 (Estimated)

PRIMARY OUTCOMES:
To characterize the epidemiological Susac's Syndrome | 9 years
  Variables collected at inclusion: Date of birth
1. To characterize the epidemiological of Susac's Syndrome | 9 years
  Variables collected at inclusion:
  • Place of birth
1. To characterize the epidemiological of Susac's Syndrome | 9 years
  • Variables collected at inclusion: Sex
1. To characterize the epidemiological of Susac's Syndrome | 9 years
  • Variables collected at inclusion : Date of first symptom
1. To characterize the epidemiological of Susac's Syndrome | 9 years
  • Variables collected at inclusion: Date of diagnosis
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at inclusion :
  • Personal medical history
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at inclusion :
  • Gynaecological history
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at inclusion :
  • Surgical history
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at inclusion :
  • Family history
2. To characterize the etiological of Susac's Syndrome | 9 years
  • Variables collected at inclusion : Previous travel and vaccination status
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at inclusion :
  • Any symptoms (flu-like illness, fever)
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at each visit :
  • - Weight in kilograms
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at each visit :
  • - Tobacco consumption
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at each visit :
  • - Use of oestroprogestogenic contraception
2. To characterize the etiological of Susac's Syndrome | 9 years
  Variables collected at each visit :
  • - Alcohol consumption
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset : Headache
3. To characterize the clinical of Susac's Syndrome | 9 years
  Neurology: Neurological symptoms: present / absent / date of onset :
  • Sensory disturbance
3. To characterize the clinical of Susac's Syndrome | 9 years
  Neurology: Neurological symptoms: present / absent / date of onset :
  • Motor deficit
3. To characterize the clinical of Susac's Syndrome | 9 years
  Neurology: Neurological symptoms: present / absent / date of onset :
  • Osteotendinous pyramidal reflexes
3. To characterize the clinical of Susac's Syndrome | 9 years
  Neurology: Neurological symptoms: present / absent / date of onset :
  • Babinski sign
3. To characterize the clinical of Susac's Syndrome | 9 years
  Neurology: Neurological symptoms: present / absent / date of onset :
  • Hoffman's sign
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Tact sensitivity disorder
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Thermoal sensitivity deficit
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  Proprioceptive disorder :
  • If yes, specify :
  * Ataxia
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  Proprioceptive disorder :
  • If yes, specify :
  * Anomaly of the sense of position of the big toe
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Paresthesias
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Encephalopathy, If yes, specify the signs present:
  * Confusion
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Encephalopathy, If yes, specify the signs present:
  * Obnubilation
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Encephalopathy, If yes, specify the signs present:
  * Coma
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Encephalopathy, If yes, specify the signs present:
  * Agitation
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Encephalopathy, If yes, specify the signs present:
  * Temporo-spatial disorientation
3. To characterize the clinical of Susac's Syndrome | 9 years
  1) Neurology: Neurological symptoms: present / absent / date of onset :
  • Encephalopathy, If yes, specify the signs present:
  * Fluctuating memory disorders
3. To characterize the clinical of Susac's Syndrome | 9 years
  • Any sequelae : Results of neurocognitive assessment : BREF
3. To characterize the clinical of Susac's Syndrome | 9 years
  Any sequelae : • Results of neurocognitive assessment: MMS
3. To characterize the clinical of Susac's Syndrome | 9 years
  Any sequelae : For mood disorders and quality of life: DSMIV criteria for depression
3. To characterize the clinical of Susac's Syndrome | 9 years
  Any sequelae : For mood disorders and quality of life: SF36
3. To characterize the clinical of Susac's Syndrome | 9 years
  Any sequelae : • For disability : Barthel Index
3. To characterize the clinical of Susac's Syndrome | 9 years
  • Any sequelae : For disability : Rankin score
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophthalmology
  • Ophthalmological examination results : Fundus
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophthalmology
  • Ophthalmological examination results : Visual field
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophthalmology
  • Ophthalmological examination results : o Angiography
3. To characterize the clinical of Susac's Syndrome | 9 years
  • Ophthalmology Ophthalmological symptoms: scotoma
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophthalmology : Ophthalmological symptoms: decrease in visual acuity
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophtalmology : Evolution of retinal arterial occlusions: improvement
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophthalmology : Evolution of retinal arterial occlusions: stability
3. To characterize the clinical of Susac's Syndrome | 9 years
  Ophthalmology : Evolution of retinal arterial occlusions: worsening
3. To characterize the clinical of Susac's Syndrome | 9 years
  • Ophthalmology : Sequelae
3. To characterize the clinical of Susac's Syndrome | 9 years
  ENT :
  * Cochlear symptoms: vertigo, tinnitus, ataxia, hearing loss
3. To characterize the clinical of Susac's Syndrome | 9 years
  ENT:
  • Audiogram results
3. To characterize the clinical of Susac's Syndrome | 9 years
  ENT
  • Results of vestibular examinations
3. To characterize the clinical of Susac's Syndrome | 9 years
  ENT
  • Course of deafness: improvement, stability, worsening
3. To characterize the clinical of Susac's Syndrome | 9 years
  ENT :
  • Possible sequelae (functional discomfort, psycho-social repercussions, follow-up audiograms)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Sacre, MD, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France